CLINICAL TRIAL: NCT05487027
Title: Can Work be Organized to Become More Health Promoting for Employees in Home Care Services?
Acronym: GoldiCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other); Trondheim Kommune (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 315556
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Occupational Exposure; Musculoskeletal Pain; Work-related Injury; Low Back Pain; Shoulder Pain; Neck Pain
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain; Shoulder Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: Individuals are grouped in clusters, where the clusters are the home care units in Trondheim. Half of the units will be randomized to control, half will be randomized to intervention. All units will be randomized at the same time.
Masking Description: No masking will be possible as the home care units will have an integral part in applying the intervention. The investigators will need to have control over the units in intervention arm as they may need to assist in the early stages of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm will have no intervention or instructions from researchers. Participants in this arm will perform their work planning as normal.
- Intervention (Experimental): Introduce a deliberate variation between workers in how much they care for physically strenuous users. Some workers may receive more strenuous work compared to before, some less.
  Interventions: Behavioral: Goldilocks work principle

INTERVENTIONS:
Behavioral: Goldilocks work principle — Using the Goldilocks work principle we have tried to find the "just right" distribution of physical strain in the home care sector. This is an intervention to test if it possible to distribute the physical strain experienced in the home care sector in a way that may be more health promoting for the workers.
  Arms: Intervention

SUMMARY:
This is a two-group, cluster randomized controlled trial designed to assess a health promoting intervention in the home care sector. The intervention aims to evenly distribute the patients requiring high levels of demanding care across all workers on the units, which may lower the working strain and thus the incidence of musculoskeletal pain. The two groups in the study will be a control group and an intervention group. The intervention will last for approximately 4 months.

DETAILED DESCRIPTION:
This is a two-group cluster randomized controlled trial to compare an organizational intervention to control. The home care units will be treated as clusters to avoid contamination within units.

Control group: No intervention, their work will continue as usual without any instructions from researchers.

Intervention group: The intervention will consist of the operational managers distributing the physically strenuous shifts evenly between the workers in each home care unit. This will be achieved using a tool developed in Microsoft Excel which gives an overview over how much strain we expect each shift to have and gives a score on how well the operational manager distributes the strain between employees.

The intervention will last for approximately 4 months, depending on duration of pre and post measurements.

ELIGIBILITY:
Inclusion Criteria:

* Home care worker in one of the included home care units in Trondheim municipality.
* More than or equal to 50% working position at the home care unit.

Exclusion Criteria:

* Physically incapable of performing day to day tasks.
* Any illness during the measurement week
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Between group changes in musculoskeletal pain in the neck and shoulder from pre to post measurement | 7 days during baseline measurements, 7 days during post measurements
  The workers will rate their musculoskeletal pain in the neck and shoulder area after each working day for a week. The measurement will be repeated at the end of the intervention to assess any changes in the experience of musculoskeletal pain. The question assessing musculoskeletal pain in shoulder and neck area is phrased as "How much pain did you have in your shoulder/neck at the end of this working day?" (Translated from Norwegian).
in musculoskeletal pain in the lower back from pre to post measurement | 7 days during baseline measurements, 7 days during post measurements
  The workers will rate their musculoskeletal pain in the lower back after each working day for one week. The measurement will be repeated at the end of the intervention to assess any changes in the experience of musculoskeletal pain. The question assessing musculoskeletal pain in the lower back area is phrased as "how much pain did you have in your lower back at the end of the working day?" (Translated from Norwegian).

SECONDARY OUTCOMES:
Between group changes in the composition of time spent standing, arms elevated and trunk inclined | 7 days during baseline measurements, 7 days during post measurements
  The difference in physical behavior composition from baseline measurements to post measurements between control and intervention group. The specific variables will be time spent standing, arms elevated, and trunk inclined.
Between group changes in fatigue at end of shift | 7 days during baseline measurements, 7 days during post measurements
  The difference between intervention and control group from pre- to post-measurements in how fatigued the workers were at the end of the shift.

CONTACTS AND LOCATIONS:
Locations (11):
- Norway (11):
  - Bergheim hjemmetjeneste, Trondheim, Trøndelag
  - Heimdal Hjemmetjeneste, Trondheim, Trøndelag
  - Klæbu hjemmetjeneste, Trondheim, Trøndelag
  - Lade hjemmetjeneste, Trondheim, Trøndelag
  - Nidarvoll hjemmetjeneste, Trondheim, Trøndelag
  - Nidelven hjemmetjeneste, Trondheim, Trøndelag
  - Saupstad hjemmetjeneste, Trondheim, Trøndelag
  - Spongdal hjemmetjeneste, Trondheim, Trøndelag
  - Strinda Hjemmetjeneste, Trondheim, Trøndelag
  - Strindheim hjemmetjeneste, Trondheim, Trøndelag
  - Valentinlyst hjemmetjeneste, Trondheim, Trøndelag

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers in my research group but not with any databases or researchers from other groups.

REFERENCES:
- [Derived] Lohne FK, Fimland MS, Palarea-Albaladejo J, Mathiassen SE, Holtermann A, Redzovic S. Can home care work be organized to promote musculoskeletal health for workers? Results from the GoldiCare cluster randomized controlled trial. BMC Health Serv Res. 2025 Jan 7;25(1):41. doi: 10.1186/s12913-024-12133-2. PMID 39773460
- [Derived] Lohne FK, Fimland MS, Holtermann A, Mathiassen SE, Fischer H, Gellein TM, Redzovic S. Can home care work be organized to promote musculoskeletal health for workers? Study protocol for the Norwegian GoldiCare cluster randomized controlled trial. BMC Health Serv Res. 2022 Dec 7;22(1):1490. doi: 10.1186/s12913-022-08916-0. PMID 36476502